CLINICAL TRIAL: NCT06700850
Title: An Open-label, Prospective, Comparative Human Participant Study to Evaluate the Clinically Acceptable Dressing Presence and Conformability Properties of Prototype Non-medicated Multilayer Foam Dressings Compared to Established Medical Devices
Brief Title: Human Participant Study of Prototype Non-medicated Multilayer Foam Dressings on Intact Skin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Smith & Nephew, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HVS2312; CIV-24-03-046336 (Other: EUDAMED)
Record Dates: First submitted 2024-11-08; First posted 2024-11-22 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2024-11

CONDITIONS: Healthy
Keywords: Foam dressing; healthy volunteers; intact skin; wear-time

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Prototype dressing (rectangle) vs Marketed dressing (rectangle) on knees (Other): Each participant will receive a comparison pair Prototype dressing (rectangle) vs Marketed dressing (rectangle) applied to knees (one dressing per knee). Each dressing of the comparison pair will be randomised to either the right or left knee in a 1:1 ratio.
  Interventions: Device: Prototype dressing rectangle; Device: Marketed dressing rectangle
- Prototype dressing (square) vs Marketed dressing (square) on thighs (Other): Each participant will receive a comparison pair Prototype dressing (square) vs Marketed dressing (square) applied to thighs (one dressing per thigh). Each dressing of the comparison pair will be randomised to either the right or left thigh in a 1:1 ratio.
  Interventions: Device: Prototype dressing square; Device: Marketed dressing square

INTERVENTIONS:
Device: Prototype dressing rectangle — Prototype multilayer foam wound dressing with polyurethane, cellulose, superabsorbent polymer, silicone adhesive, acrylic adhesive. LDPE (Low Density Polyethylene). Size: 30x10cm. Topical application. Single use.
  Arms: Prototype dressing (rectangle) vs Marketed dressing (rectangle) on knees
Device: Marketed dressing rectangle — CE marked multilayer foam wound dressing with silicone, polyurethane, viscose, polyester, polyolefins, polyacrylate and superabsorbent acrylate fibres. Size: 30x10cm. Topical application. Single use
  Arms: Prototype dressing (rectangle) vs Marketed dressing (rectangle) on knees
Device: Prototype dressing square — Prototype multilayer foam wound dressing with polyurethane, cellulose, superabsorbent polymer, silicone adhesive, acrylic adhesive. LDPE (Low Density Polyethylene). Size: 7.5x7.5cm. Topical application. Single use.
  Arms: Prototype dressing (square) vs Marketed dressing (square) on thighs
Device: Marketed dressing square — CE marked multilayer foam wound dressing with silicone, polyurethane, viscose, polyester, polyolefins, polyacrylate and superabsorbent acrylate fibres. Size: 7.5x7.5cm. Topical application. Single use.
  Arms: Prototype dressing (square) vs Marketed dressing (square) on thighs

SUMMARY:
The purpose of this study is to evaluate two new prototype non-medicated multilayer foam dressings on healthy, intact skin.

The study will find out how well two new prototype dressings stay in place as well as other dressing performance and safety factors when compared to corresponding, marketed dressings with a similar intended use profile and shape.

The study will compare:

1. Prototype dressing (rectangle) vs Marketed dressing (rectangle) on the knee.
2. Prototype dressing (square) vs Marketed dressing (square) on the thigh.

The main aim of the study is to show that the new prototype dressings are not worse than the established marketed comparison dressings in terms of staying in place on human participants at 7 days.

Dressings will have successfully stayed in place if the dressing edges have not lifted to reach the pad, and the pad is not exposed in any way.

Additional data will be collected to further support product performance up to 7 days, including safety information and potential device issues.

DETAILED DESCRIPTION:
This is a single-centre, prospective, open-label, comparative, interventional study with intra-individual comparison.

Four different dressings (two prototype investigational medical devices (IMDs) and two comparators) will be investigated, with each participant receiving all dressings. The dressings will be divided into two comparison pairs:

(i) Prototype dressing (rectangle) vs Marketed dressing (rectangle) (ii) Prototype dressing (square) vs Marketed dressing (square)

Comparison pair (i) will be applied to the knees (one dressing per knee) and comparison pair (ii) will be applied to the thighs (one dressing per thigh). The two dressing in each comparison pair will be randomised to either the right or left knee / thigh in a 1:1 ratio.

120 participants will be recruited into this study at a single, Germany-based site. The sample size accounts for the required 105 evaluable participants and approximately 10% lost to follow-up rate. Participants will be in good general health and have intact skin.

Duration of the study will be 7-14 days, with participants attending 5 site visits. Screening can be completed on Day 0 or at a separate visit up to 7 days prior to Day 0. Dressings will be worn by participants for up to 7 days.

A screening visit will be completed Day -7 to Day 0 to assess participant eligibility and to perform informed consent. Objective and subjective assessments during visits will evaluate dressing performance and conformability properties. On Day 0, dressings will be applied after appropriate skin assessments. On Day 1, 3 and 7, assessments will include acceptable dressing presence, retention, pad integrity, pad lift, border lift, and dressing comfort. On Day 1, the assessments will be performed before and after a physiotherapy regime to evaluate dressing performance following mobilization of the leg/knee joint. On Day 7 or at dressing removal, additional assessments will include adhesive offset on skin, ease of removal and pain on removal. At each visit, photographs of the dressings will be taken. Furthermore, at each visit the skin at the application site will be assessed for any Adverse Events (AE) and the dressings assessed for Device Deficiencies.

ELIGIBILITY:
Inclusion Criteria:

* Participant is capable of providing informed consent
* Participant is willing and able to make all required study visits
* Aged 22-70 years at the time of signing the informed consent*
* Participant must be in good health, as determined by the Investigator, based on medical evaluation, including medical history and skin application site assessment (healthy intact skin at or near any of the dressing application sites)
* Participant is willing not to use cosmetic or medicinal lotions, creams, ointments and anything else which may interfere with dressing adhesion at dressing application sites for the duration of the study from 24 hours before dressing application on Day 0.
* Participant is willing to have excess hair removed from the dressing application sites
* Participant is willing to avoid immersing the dressings in water (no swimming or bathing) for the duration of the study

Footnote:

* at least 10% of participants are aged >55 years

Exclusion Criteria:

* Female participant who is pregnant, or lactating.
* Participant has a known sensitivity to any of the study products, materials or ancillary product or components.
* Known skin sensitivity or allergies to adhesives, skin wipes, soap, surgical first-aid dressings, natural rubber or rubber latex, etc.
* Participants with a current active skin disease (e.g., eczema, psoriasis, or severe dermatoporosis), sunburn or skin peeling at the dressing application sites.
* Participants with a medical condition which may interfere with their perception of pain (such as diabetes, small-fibre neuropathy, allodynia, hyperalgesia etc.).
* Heavy smokers (e.g. >20 cigarettes (~1 pack) a day over the last 10 years) whose pain perception may have been affected through smoking.
* Participants with any skin features near any of the dressing application sites that could be identifiable/may interfere with skin assessments (e.g. tattoos/distinctive markings or scars/keloids).
* Participants diagnosed with hyperhidrosis or who self-report their normal sweating level to be severe as determined by the Sweating Severity Self-Assessment (SSSA) at screening (e.g. mild, moderate, severe).
* Participants not willing to refrain from the use of pain relief medication on assessment days (0, 3, 5 and 7) and in the case of certain medications, 24 hours before assessments.
* Participants unwilling to refrain from activities which may directly affect the dressing, dressing application sites or assessments (such as undergoing planned scanning procedures, e.g., X-ray, magnetic resonance imaging (MRI) and computed tomography (CT) scanning; exposure to airport scanners or devices emitting radio waves; exposure to atypical conditions of pressure, humidity and temperature; immersing the dressing in water e.g. bathing / swimming / cleaning the dressing application sites; using a sauna; undertaking strenuous physical activity like aerobics, running, cycling, heavy labor etc.; using lotions/creams/ointments etc. at the dressing application sites; excessively exposing the dressing application sites to the sun (e.g. sunbathing for >1 hour); wearing tightly fitting clothes which could affect the dressings.
* Individuals who have participated in a clinical study in the last 7 days, using the same dressing application sites.
* Participants with poor compliance and / or poor willingness to co-operate.
* Individuals who should not participate in the clinical investigation for any other reason (including the taking of certain medications and with respect to the physiotherapy session) as judged by the Investigator.
* Individuals who are inmates in psychiatric wards, prison or state institutions, or any individuals otherwise regarded as vulnerable (as per ISO 14155 Section 3.55).
* Employees of the investigation sites directly involved in this clinical investigation or employees of the sponsor's company.

Ages: 22 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2024-10-28 (Actual); Primary Completion 2025-01-21 (Actual); Study Completion 2025-01-21 (Actual)

PRIMARY OUTCOMES:
Acceptable Dressing Presence at Day 7 | Day 7
  Acceptable dressing presence determined by a yes/no assessment at day 7, with a 'yes' response defined as the dressing is in place with no border lift reaching the pad and no pad exposure.

SECONDARY OUTCOMES:
Acceptable Dressing Presence at Day 1 and Day 3 | Day 1 and Day 3
  Acceptable dressing presence determined by a yes/no assessment at Day 1 and 3, with a 'yes' response defined as the dressing is in place with no border lift reaching the pad and no pad exposure.
Presence of Dressing | Day 1, Day 3 and Day 7
  Dressing presence determined at Day 1, 3 and 7 by response to the question "Is the dressing in place?" (yes/no).
Pad Integrity | Day 1, Day 3 and Day 7
  Changes to the integrity of the dressing pad (e.g., bunching, folding, ridges) assessed at Day 1, 3 and 7 by one of the following categories:
  1. 0% (no change)
  2. 1-25%
  3. 26%-50%
  4. 51%-75%
  5. 76-100%
  6. Dressing missing
Pad Lift | Day 1, Day 3 and Day 7
  Lift of the dressing pad assessed at Day 1, 3 and 7 to determine the extent of pad area lifted and no longer adhered to the participant's skin by one of the following percentage categories:
  1. 0% (no lift)
  2. 1-25%
  3. 26%-50%
  4. 51%-75%
  5. 76-100%
  6. Dressing missing
Border Lift | Day 1, Day 3 and Day 7
  Lift of the dressing border assessed at Day 1, 3 and 7 to determine the extent of the border area lifted and no longer adhered to the participant's skin by one of the following percentage categories:
  1. 0% (no lift)
  2. 1-25%
  3. 26%-50%
  4. 51%-75%
  5. 76-100%
  6. Dressing missing
Dressing Comfort | Day 1, Day 3 and Day 7
  Dressing comfort assessed at Day 1, 3 and 7 by the participant's answer to the question "was the dressing comfortable during wear?" from one of the following responses:
  1. Yes
  2. No
  3. Dressing missing

CONTACTS AND LOCATIONS:
Overall Officials: Kirstin Deuble-Bente, Principal Investigator — SGS proderm
Locations (1):
- SGS proderm, Schenefeld, Schleswig-Holstein, Germany

IPD SHARING:
Plan to Share IPD: No